CLINICAL TRIAL: NCT03084939
Title: A Randomized, Multicenter, Phase III Open-Label Study of the Efficacy and Safety of Trastuzumab Emtansine Versus Lapatinib Plus Capecitabine in Chinese Patients With HER2-Positive Locally Advanced or Metastatic Breast Cancer Who Have Received Prior Trastuzumab-Based Therapy
Brief Title: Efficacy and Safety of Trastuzumab Emtansine in Chinese Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO29919
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trastuzumab Emtansine (Experimental): Participants with HER2-positive, unresectable LABC or MBC who have experienced disease progression after treatment with trastuzumab and a taxane will be treated with trastuzumab emtansine. Participants may continue to receive study treatment until disease progression (as assessed by the investigator), unmanageable toxicity, or study termination by the Sponsor.
  Interventions: Biological: Trastuzumab Emtansine
- Control (lapatinib + capecitabine) (Active Comparator): Participants with HER2-positive, unresectable LABC or MBC who have experienced disease progression after treatment with trastuzumab and a taxane will be treated with lapatinib plus capecitabine. Participants may continue to receive study treatment until disease progression (as assessed by the investigator), unmanageable toxicity, or study termination by the Sponsor.
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Biological: Trastuzumab Emtansine — Trastuzumab emtansine 3.6 milligrams per kilogram (mg/kg) was administered intravenously on Day 1 of each 21-day cycle.
  Other Names: Kadcyla
  Arms: Trastuzumab Emtansine
Drug: Lapatinib — Lapatinib 1250 mg was administered orally once per day of each 21-day cycle.
  Arms: Control (lapatinib + capecitabine)
Drug: Capecitabine — Capecitabine 1000 milligrams per square meter (mg/m^2) was administered orally twice daily on Days 1-14 of each 21-day cycle.
  Arms: Control (lapatinib + capecitabine)

SUMMARY:
This is a Phase III, randomized, multicenter, two-arm, open-label study designed to evaluate the safety and efficacy of trastuzumab emtansine compared with that of lapatinib + capecitabine in Chinese participants with HER2-positive, unresectable locally advanced breast cancer (LABC) or metastatic breast cancer (MBC) who have received prior trastuzumab-based therapy. A total of approximately 350 participants will be enrolled in China. The study will consist of 2 stages. Stage 1: Eligible participants will be randomized in a 3:1 ratio to receive either trastuzumab emtansine or control (lapatinib + capecitabine). Stage 2: After Stage 1 is recruited, eligible patients will be enrolled to receive trastuzumab emtansine only.

ELIGIBILITY:
Inclusion Criteria:

* Aged >/= 18 years
* Prospective centrally assessed HER2-positive disease (i.e., immunohistochemistry [IHC] 3+ and/or gene amplified [HER2 to Chromosome 17 [CEP 17] ratio >/= 2]) by in situ hybridization (ISH) through use of archival paraffin-embedded tumor tissue
* Histologically or cytologically confirmed invasive breast cancer (BC): incurable, unresectable LABC previously treated with multimodality therapy or MBC
* Prior treatment for BC in the adjuvant, unresectable locally advanced or metastatic setting must include both: a taxane, alone or in combination with another agent, and trastuzumab, alone or in combination with another agent in the adjuvant, unresectable locally advanced or metastatic setting
* Documented progression of incurable, unresectable LABC or MBC, defined by the investigator: progression must occur during or after most recent treatment for LABC or MBC or within 6 months after completing adjuvant therapy
* Measurable and/or non-measurable disease, according the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 definition: CNS-only disease excluded
* Left ventricular ejection fraction (LVEF) >/=50% by either echocardiogram or multiple-gated acquisition
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate organ function evidenced by laboratory results within 30 days prior to randomization
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study drug
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures (use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year) and agreement to refrain from donating sperm during the treatment period and for at least 7 months after the last dose of study drug

Exclusion Criteria:

* History of treatment with trastuzumab emtansine
* Prior treatment with lapatinib or capecitabine
* Peripheral neuropathy of Grade >/= 3 per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0)
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, synchronous or previously diagnosed HER2-positive BC, or cancers with a similar curative outcome as those mentioned above
* History of receiving any anti-cancer drug/biologic or investigational treatment within 21 days prior to randomization, except hormone therapy which can be given up to 7 days prior to randomization
* History of radiation therapy within 14 days before randomization
* Brain metastases that are untreated, symptomatic, progressive, or require therapy such as radiation, surgery or corticosteroid therapy to control symptoms from brain metastases within 30 days before randomization
* History of exposure to cumulative doses of anthracyclines: Doxorubicin > 500 milligrams per square meter (mg/m^2), Epirubucin > 720 mg/m^2, Mitoxantrone > 120 mg/m^2
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
* Pregnancy or lactation
* Currently known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Presence of conditions that could affect gastrointestinal absorption
* History of intolerance (including Grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins
* Known hypersensitivity to 5-fluorouracil or known dihydropyrimidine dehydrogenase deficiency
* Current treatment with sorivudine or its chemically related analogs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 17 months
  PFS is defined as the time from randomization to the first occurrence of disease progression as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) Version (v1.1), or death from any cause during the study, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 millimeter (mm) taking as reference the smallest sum during the study including baseline or the appearance of one or more new lesions. Tumor assessments will be performed with computed tomography (CT) or magnetic resonance imaging (MRI) scans.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 29 months
  ORR is defined as percentage of participants with partial response (PR) or complete response (CR) determined on the basis of investigator assessments with the use of RECIST v1.1. CR: disappearance of all target lesions; PR: >/= 30% decrease in the sum of the longest diameters of target lesions taking as reference baseline sum diameters; Objective Response Rate (OR) = CR + PR. Tumor assessments will be performed with CT or MRI scans.
Duration of Response (DOR) | Up to approximately 29 months
  DOR is defined as as the time from the date of initial confirmed PR or CR to the date of disease progression or death within the study. CR: disappearance of all target lesions; PR: >/= 30% decrease in the sum of the longest diameters of target lesions taking as reference baseline sum diameters. Disease progression was defined according to RECIST, v1.1 as at least a 20% increase in the sum of diameters of target lesions with an absolute increase of at least 5 mm or the appearance of one or more new lesions. Tumor assessments will be performed with CT or MRI scans.
Overall Survival (OS) | When at least 100 (50%) death events are observed from participants in Stage 1
  OS is defined as the time from the date of randomization to the date of death from any cause.
Number of Participants with Adverse Events | Up to approximately 56 months
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Serum Concentration of Trastuzumab Emtansine Conjugate | Pre-dose and 15-30 minutes after dose on Day 1 of each 21-day cycle during Cycles 1-4 and at completion/early termination visit (up to approximately 56 months)
  Concentration of trastuzumab emtansine conjugate will be measured in serum from participants, who received trastuzumab emtansine.
Plasma Concentration of N2'-deacetyl-N2'-(3-mercapto-1-oxopropyl)-maytansine (DM1) | Pre-dose on Day 1 of Cycle 1, 15-30 minutes after dose on Day 1 of each 21-day cycle during Cycles 1-4
  Concentration of the analyte DM1 will be measured in plasma from participants, who received trastuzumab emtansine.
Serum Concentration of Total Trastuzumab | Pre-dose and 15-30 minutes after dose on Day 1 of each 21-day cycle during Cycles 1-4
  Concentration of total trastuzumab will be measured in serum from participants, who received trastuzumab emtansine.
Percentage of Participants with Anti-therapeutic Antibodies (ATA) to Trastuzumab Emtansine | Pre-dose on Day 1 of Cycle 1 and Day 1 of Cycle 4, at completion/early termination visit and 3 months after last dose of trastuzumab emtansine (up to approximately 56 months)
  ATA to trastuzumab emtansine were measured in serum of participants, who received trastuzumab emtansine.
Patient-reported Outcome: Percentage of Participants with Clinically Significant Deterioration | Day 1 (prior to any study procedures or discussion of test results) of Cycle 1 (21 days) and every two cycles thereafter until treatment discontinuation and at the completion/early termination visit (up to approximately 56 months)
  The patient-reported outcome of clinically significant deterioration in physical well-being, functional well-being, and breast cancer symptoms will be determined by a decrease of >/= 5 points from baseline on the Performance/Functional/Breast (PFB) Trial Outcome Index (TOI) score of the Functional Assessment of Cancer Therapy-Breast (FACT-B, Version 4) questionnaire in female participants only. Reported here is the percentage of participants with clinically significant deterioration.
Patient-reported Outcome: Time to Clinically Significant Deterioration | Day 1 (prior to any study procedures or discussion of test results) of Cycle 1 (21 days) and every two cycles thereafter until treatment discontinuation (up to approximately 56 months)
  The patient-reported outcome of clinically significant deterioration in physical well-being, functional well-being, and breast cancer symptoms will be determined by a decrease of >/= 5 points from baseline on the PFB TOI score of the FACT-B, Version 4 questionnaire in female participants only. Reported here is the time to clinically significant deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- China (18):
  - Beijing Hospital, Beijing
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - Beijing Cancer Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Changzhou First People's Hospital, Changzhou
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - The Second Affiliated Hospital of Zhejiang University College, Hangzhou
  - Zhejiang Cancer Hospital; Zhejiang Cancer Hospital cancer department, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Province Hospital, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning cancer Hospital & Institute, Shenyang
  - Tianjin Cancer Hospital, Tianjin
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an

REFERENCES:
- [Derived] Wang X, Li W, Yin Y, Tong Z, Zhang Q, Zheng H, Shao Z, Li H, Yang J, Feng J, Wu F, Lamour F, Restuccia E, Jiang Z. Primary results of ELAINA: a randomized, multicenter, open-label, phase III study of the efficacy and safety of trastuzumab emtansine vs. lapatinib plus capecitabine in Chinese patients with HER2-positive locally advanced or metastatic breast cancer who have received prior trastuzumab-based therapy. Transl Breast Cancer Res. 2023 Jan 31;4:3. doi: 10.21037/tbcr-23-2. eCollection 2023. PMID 38751488